CLINICAL TRIAL: NCT06021834
Title: Effect of Physical Rehabilitation on Cardiorespiratory Parameters, Postural Balance and Sociopsychological and Cognitive Variables in Patients With Parkinson's Disease
Brief Title: Effect of Physical Rehabilitation in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Ghazoua Nafti, Principal Investigator Ghazoua NAFTI, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Faculté de Médecine de Sousse
Record Dates: First submitted 2023-05-30; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: "Parkinson Disease"; "cognitive function"; "postural balance"; "physical rehabilitation"
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group will be invited to attend the program three times per week and will engage in an endurance training program
  Interventions: Other: rehabilitation
- experimental group (Experimental): the experimental group will be invited to attend the program three times per week and will participate in a combined endurance training and cognitive training program.
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — The subjects will be invited to attend the program three times per week.

SUMMARY:
This is a prospective study. The aim of this study is to investigate the effect of exercise retraining on cardiorespiratory parameters, postural balance, sociopsychological variables, and cognitive function in subjects with Parkinson's disease.

There will be two measurement sessions, one pre-intervention and one post-intervention (measuring cardiorespiratory parameters, evaluating dynamic and static postural balance, and assessing cognitive function).

DETAILED DESCRIPTION:
this is a 12-week prospective study with the theme that I wish to develop in this context entitled "the effect of exercise retraining on cardiorespiratory parameters, postural balance, sociopsychological variables, and cognitive function in subjects with Parkinson's disease".

There will be two measurement sessions, one pre-intervention and one post-intervention (measuring cardiorespiratory parameters, evaluating dynamic and static postural balance, and assessing cognitive function).

The recruited subjects will be randomly assigned to two groups: a control group and an experimental group. The subjects will be invited to attend the program three times per week.

The control group will engage in an endurance training program, while the experimental group will participate in a combined endurance training and cognitive training program

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease according to the Movement Disorder Society (MDS) 2015 criteria.
* Mild to moderate stage according to the Hoehn and Yahr scale.
* No hearing or visual impairments that could hinder the integration and implementation of the rehabilitation protocol.
* Has the ability to communicate and walk.
* Patient has been stable on treatment for 3 months.

Exclusion Criteria:

* A contraindication to engaging in cardiovascular physical activity
* A Montreal Cognitive Assessment score (MoCA ) of less than 24.
* A current psychiatric disorder that could make it difficult or dangerous to adhere to the research protocol.
* Musculoskeletal impairments or excessive pain in any joint that could limit participation in an exercise program.
* Treatment with sedative medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-08 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Parameters | There will be two measurement sessions, one pre-intervention and one post-intervention (After 12 week for each patient)
  Cardiorespiratory Parameters will be assessed using the six-minute walk test (6MWT).
Postural Balance | There will be two measurement sessions, one pre-intervention and one post-intervention (After 12 week for each patient)
  Postural balance will be assessed using the Timed Up and Go test (TUG) and stabilometry platform
Depression | There will be two measurement sessions, one pre-intervention and one post-intervention (After 12 week for each patient)
  The depression variable will be assessed through Beck Depression Inventory-II .
Cognitive Function | There will be two measurement sessions, one pre-intervention and one post-intervention (After 12 week for each patient)
  Cognitive function will be evaluated using the Montreal Cognitive Assessment score (MoCA) .

SECONDARY OUTCOMES:
Strength | There will be two measurement sessions, one pre-intervention and one post-intervention (After 12 week for each patient)
  handgrip test, Functional Reach Test, Five time to sit and stand test